CLINICAL TRIAL: NCT04784156
Title: The Use of a Sustained Dynamic Compression Intramedullary Nail for Subtalar Arthrodesis
Brief Title: Use of a Sustained Dynamic Compression Intramedullary Nail for Subtalar Arthrodesis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: MedShape, Inc (Industry)
Collaborators: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00104048
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-03

CONDITIONS: Foot Arthritis
Keywords: Subtalar Arthrodesis; Intramedullary Nail; Sustained Dynamic Compression; Internal Fixation
MeSH Terms: interventions — Arthrodesis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- All study patients: All study patients will be in one group.
  Interventions:
  Procedure: Subtalar (Talocalcaneal) arthrodesis Device: DynaNail Mini
  Interventions: Procedure: Subtalar (Talocalcaneal) Arthrodesis; Device: DynaNail Mini

INTERVENTIONS:
Procedure: Subtalar (Talocalcaneal) Arthrodesis — Subtalar (Talocalcaneal) arthrodesis with a novel sustained dynamic compression intramedullary nail
Device: DynaNail Mini — Utilization of a novel sustained dynamic compression pseudoelastic intramedullary nail

SUMMARY:
The purpose of this study is to determine the clinical efficacy of a novel dynamic sustained compression intramedullary nail for subtalar (talocalcaneal) arthrodesis.

DETAILED DESCRIPTION:
This proposal is a collaborative effort between MedShape and the Medical University of South Carolina. This is a prospective investigation to assess the clinical outcomes of patients with a subtalar arthrodesis with the Sustained Dynamic Compression Intramedullary Nail (DynaNail Mini). The study plan is to enroll 60 patients.

Patients with end-stage talocalcaneal (subtalar) joint arthritis from any etiology will be asked to enroll in the study. After informed consent, the patients will be asked to complete the following patient reported outcomes questionnaires as part of the Surgical Outcomes System (SOS) Global Registry: Visual Analog Scale (VAS) for pain, Veterans RAND 12 Item Health Survey for function, Foot Function Index - Revised for function and pain, the Foot and Ankle Ability Measure (FAAM) for function, and the American Orthopaedic Foot and Ankle Society (AOFAS) scales for pain, function, and alignment. After informed consent, they will then be scheduled for surgery in a routine fashion.

The following surgical procedure is standard of care. The surgical procedure will involve subtalar (talocalcaneal) joint preparation through a lateral approach. The use of supplemental bone graft is at the discretion of the treating surgeon but must be documented. The MedShape DynaNail Mini will then be inserted according to the manufacturer's technique. The patient will be placed in a short leg splint and kept non-weight bearing. The patient will be discharged from the hospital when medically ready.

The patient will return to clinic for visits at the following intervals after surgery: 6 (+/- 1) weeks, 14 (+/- 1) weeks, 6 months (+/- 2 weeks), and 12 months (+/- 2 weeks). At each of these time points, the same SOS patient specific outcome questionnaires will be administered. 3-view X-rays will be taken at each of these visits to assess the amount of travel of the Mini compressive element. At 15 (+/- 1) weeks post-op, a CT scan will be obtained to assess healing. Additionally, a radiographic and clinical follow-up form will be filled out at each of the following follow-up visits: 6 weeks, 14 weeks, 6 months, and 1 year.

Patients will be identified in the clinic by an attending orthopaedic foot and ankle surgeon or his physician assistant based on clinical exam and radiographic findings. Inclusion criteria include anyone over age 18 who has end-stage subtalar arthritis and has failed nonoperative management. Typically, these patients have multiple medical comorbidities and therefore the exclusion criteria will be patients who are not healthy enough to undergo surgery. Additional exclusion criteria include non-English speakers, and patients that are blind, illiterate, or are prisoners. Additionally, pregnant women will be excluded. Patients of all racial, religious, and cultural backgrounds will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

* End-stage talocalcaneal (subtalar) joint arthritis from any etiology will be eligible to enroll in the study
* Meets indications for subtalar arthrodesis to receive the DynaNail Mini implant
* Able to understand the requirements of the study, provide a written consent, and willing to comply with the study protocol
* 18 years of age or older

Exclusion Criteria:

* Investigator determines that the subject is unlikely to comply with the requirements of the study
* Non-English speaker
* Blind
* Illiterate
* Prisoner
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified in the clinic by an attending orthopaedic foot and ankle surgeon or his physician assistant based on clinical exam and radiographic findings. Patients will be screened for eligibility by the research coordinator/ key personnel in close coordination with the surgeon.
  Patients at institute with end-stage talocalcaneal (subtalar) joint arthritis from any etiology will be eligible to enroll in the study. Frequently, subtalar arthritis is caused by trauma. Traumatic injuries have no predilection for race, religion, cultural background, etc. Therefore, all demographic groups will have access to this study and should be represented. Approximately 60 patients will be recruited for the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Fusion | From surgery up to one year post-surgery
  Joint Fusion, as measured by radiograph and CT scan

SECONDARY OUTCOMES:
VAS | Pre-Operative up to one year post-surgery
  Pain Visual Analog Scale (VAS) - Rates the intensity of pain from 0 - 10 with 10 being the worst pain possible.
Veterans RAND 12 Item Health Survey (VR-12) | Pre-Operative up to one year post-surgery
  The Veterans RAND 12 Item Health Survey (VR-12, formerly called the Veterans SF-12) was Version Date 01.27.2020 3 developed from the Veterans RAND 36 (VR-36, formerly called the Veterans SF-36), which was modified from the original Medical Outcomes Survey (MOS) SF-36. The VR-12 measures Physical functioning (PF), social functioning (SF), role limitation due to physical problems (RP), role limitation due to emotional problems (RE), mental health (MH), energy and vitality (VT), bodily pain (BP) and general perception of health (GH). Standard based scoring (sometimes called norm based scoring) is used to calculate the physical component summary (PCS) and mental component summary (MCS) for both measures. The PCS and MCS are standardized using a t-score transformation and normed to a US population at a score of 50 and a standard deviation of 10.
Revised FFI-R | Pre-Operative up to one year post-surgery
  Measures the impact of foot pathology on function in terms of pain, disability, and activity restriction. The score is a percentage. The higher the score, the greater the disability.
Foot and Ankle Ability Measure (FAAM) | Pre-Operative up to one year post-surgery
  Measures activities of daily living and sports. The final score is a percentage. The higher final score represents a higher level of physical function.
American Orthopaedic Foot and Ankle Society Scales (AOFAS) | Pre-Operative up to one year post-surgery
  Clinician-based outcome that measures foot/ankle pain, function, and alignment. The lower the score, the greater the disability. The maximum score is 100.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Gross, MD, Principal Investigator — ASSOCIATE PROFESSOR
Locations (1):
- The Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No